CLINICAL TRIAL: NCT00635622
Title: A Phase IIa Study of the Colonization Efficiency, Safety and Acceptability of LACTIN-V Administered Vaginally to Women With Bacterial Vaginosis
Brief Title: Safety and Efficacy Study of Lactobacillus Administered Vaginally in Women With Bacterial Vaginosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osel, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Peter Lee, MD, Osel, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LV-006
Record Dates: First submitted 2008-03-10; First posted 2008-03-14 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-03

CONDITIONS: Bacterial Vaginosis
Keywords: Bacterial Vaginosis; BV; UCSF; SFGH
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vaginal application of single-use applicators pre-filled with LACTIN-V (Formulation 1) at 2 x 10^9 cfu/dose. The study product will be administered once daily for 5 consecutive days, followed by once weekly application over 2 consecutive additional weeks.
  Interventions: Drug: LACTIN-V
- 2 (Placebo Comparator): Vaginal application of single-use applicators pre-filled with placebo control substance. The study product will be administered once daily for 5 consecutive days, followed by once weekly application over 2 consecutive additional weeks.
  Interventions: Drug: Placebo control substance

INTERVENTIONS:
Drug: LACTIN-V — Vaginal application of single-use applicators pre-filled with LACTIN-V (Formulation 1) at 2 x 10^9 cfu/dose or placebo control substance. The study product will be administered once daily for 5 consecutive days, followed by once weekly application over 2 consecutive additional weeks.
  Arms: 1
Drug: Placebo control substance — Vaginal application of single-use applicators pre-filled with placebo control substance. The study product will be administered once daily for 5 consecutive days, followed by once weekly application over 2 consecutive additional weeks.
  Arms: 2

SUMMARY:
This is a phase IIa clinical trial in women with bacterial vaginosis. This study will determine whether treatment with vaginal lactobacillus in combination with antibiotic therapy (metronidazole) is effective in colonizing the vagina with the lactobacillus bacteria found in normal vaginal flora.

DETAILED DESCRIPTION:
Phase IIa randomized, double blind, placebo-controlled, clinical trial of LACTIN-V at 2 x 10^9 cfu/dose versus placebo, administered vaginally with a pre-filled applicator once daily for five consecutive days followed by a weekly dose over 2 additional weeks after an initial standardized antibiotic treatment with 0.75% topical metronidazole (MetroGel). A single site will enroll 40 participants (30 randomized to LACTIN-V and 10 to placebo).

Colonization rate of Lactobacillus crispatus CTV 05 will be assessed with culture and rep-PCR.

Safety will be determined by comparing the incidence of adverse events and serious adverse events in the LACTIN-V and placebo groups as determined by clinical symptoms, physical examination, pelvic examination with colposcopy and laboratory measurements. Tolerability will be measured by percentage of subjects who discontinue study product use due to overt adverse events and percentage of subjects who adhere to complete dosing schedule. Acceptability will be assessed via a standardized questionnaire and focus group discussions.

ELIGIBILITY:
Inclusion Criteria:

* Untreated BV (asymptomatic or symptomatic) as diagnosed during the screening visit using Amsel criteria AND confirmed in the laboratory using the Nugent scoring system (Nugent Score ≥ 7).
* Otherwise healthy pre-menopausal women 18-40 years of age at date of screening.
* Regular menstrual cycles (21-35 days) or amenorrheic for at least 3 months due to use of a long acting progestin or continuous use of oral contraceptives.
* Subject is willing to insert pre-filled vaginal applicators.
* Subject is willing to be asked questions about personal medical health and sexual history.
* Normal Pap smear collected at the screening visit. If a subject's Visit 0 Pap smear result is any of the following, the person is ineligible for participation: ASC-US (atypical squamous cells of undetermined significance), AGC (atypical glandular cells), ASC-H (atypical squamous cells, cannot r/o high grade lesion), LSIL (low grade squamous intraepithelial lesions), HSIL (high grade squamous intraepithelial lesions), adenocarcinoma in situ, adenocarcinoma, squamous cell carcinoma in situ, squamous cell carcinoma or inadequate sample.
* Vaginal and cervical anatomy that in the opinion of the Investigator lends itself easily to colposcopy.
* Capable of reading and writing English and providing informed consent.
* Previous sexual experience including vaginal intercourse.
* Previous gynecological examinations.
* Currently in a mutually monogamous sexual relationship or not sexually active.
* Agree to be sexually abstinent 72 hours prior to Visit 1 (enrollment) until Visit 2 (Day 10). Also, agree to refrain from intercourse for 48 hours after the study product application on Day 12 and 19 as well as 72 hours before the last study visit on Day 28.
* Agree to abstain from the use of any other intravaginal product (i.e., contraceptive creams, gels, foams, sponges, lubricants, douches, etc.) throughout the trial period, from the time of screening until Day 28.
* Agree to abstain from using tampons throughout the trial period, from the time of screening until Day 28.
* Agree to use an adequate method of birth control for the duration of the study to avoid pregnancy. Acceptable methods include a history of tubal ligation, male partner with a vasectomy, a steroidal contraceptive (oral, patch, injectable or implantable), IUD (Paragard or Mirena), condoms or abstinence.
* Subject must have access to functioning refrigerator.

Exclusion Criteria:

* Urogenital infection at screening or within the 21 days prior to screening. This includes urinary tract infection, Trichomonas vaginalis, Neisseria gonorrhoeae, Chlamydia trachomatis or Treponema pallidum. Subjects may be re-screened at least 21 days after the respective antibiotic or antifungal therapies have been completed.
* History of recurrent genital herpes.
* Diagnosis of N. gonorrhoeae, C. trachomatis, T. pallidum or T. vaginalis on two or more occasions during the six months prior to screening.
* Pregnancy or within 2 months of last pregnancy (all subjects will have a urine pregnancy test prior to enrollment).
* Lactation.
* Vaginal or systemic antibiotic or antifungal therapy within 21 days of the Screening visit or within 30 days of Enrollment visit.
* Investigational drug use within 30 days or 10 half-lives of the drug, whichever is longer, of enrollment visit. Planned investigational drug use while participating in this study.
* Menopause.
* IUD insertion or removal within the last 3 months.
* Pelvic surgery within the last 3 months.
* Cervical cryotherapy or cervical laser within the last 3 months.
* Use of a NuvaRing® within 3 days of the screening visit or during the course of the study.
* New long-acting treatments (e.g. depot formulation including medroxyprogesterone acetate (DMPA) form of hormonal birth control). Subjects may be enrolled if stable (> 3months) on existing therapy as determined by the Principal Investigator.
* Diabetes or other significant disease or acute illness that in the Investigator's assessment could complicate the evaluation.
* Known HIV infection or positive HIV test at screening.
* Immunosuppressive drug within 60 days.
* Previous participation in a L. crispatus CTV-05 clinical study.
* Colposcopic findings at the enrollment visit involving significant deep disruption of the epithelium.
* Known allergy to any component of LACTIN-V, other significant drug allergy or to latex (condoms).
* Unavailable for follow-up visits.
* History of drug or alcohol abuse.
* At enrollment, have any social or medical condition, or psychiatric illness that, in the opinion of the Investigator, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the vaginal colonization efficiency of L. crispatus CTV-05 after vaginal administration of LACTIN-V at 2 x 10^9 cfu/dose (600 mg) daily for 5 days followed by weekly applications over 2 additional weeks | 4 weeks after intervention

SECONDARY OUTCOMES:
To evaluate the safety of L. crispatus, LACTIN-V in otherwise healthy pre-menopausal women with BV, immediately after standardized antibiotic treatment with 0.75% topical metronidazole | 10 days and 4 weeks after intervention
To evaluate the tolerability and acceptability of LACTIN-V as a powder in a pre-filled applicator | 4 weeks after intervention
To evaluate and compare vaginal flora by Gram stain before and after receipt of LACTIN-V or placebo. | 10 days and 4 weeks after intervention
To identify and compare bacteria colonizing the vagina at screening in women with bacterial vaginosis and after antibiotic and probiotic treatment. | Before intervention and 4 weeks after intervention
To measure and compare the 4 week cure rate of BV after receipt of MetroGel in women who receive LACTIN-V or placebo. | 4 weeks after intervention
To measure the rate of vaginal colonization by Candida sp. and symptomatic vaginal candidiasis after receiving LACTIN-V or placebo | 4 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Cohen, MD, MPH, Principal Investigator — University of California, San Francisco; Anke Hemmerling, MD, MPH, PhD, Study Director — University of California, San Francisco
Locations (1):
- San Francisco General Hospital (SFGH), University of California, San Francisco (UCSF), San Francisco, California, United States

REFERENCES:
- [Background] Giorgi A, Torriani S, Dellaglio F, Bo G, Stola E, Bernuzzi L. Identification of vaginal lactobacilli from asymptomatic women. Microbiologica. 1987 Oct;10(4):377-84. PMID 3695985
- [Background] Antonio MA, Hawes SE, Hillier SL. The identification of vaginal Lactobacillus species and the demographic and microbiologic characteristics of women colonized by these species. J Infect Dis. 1999 Dec;180(6):1950-6. doi: 10.1086/315109. PMID 10558952
- [Background] Antonio MA, Hillier SL. DNA fingerprinting of Lactobacillus crispatus strain CTV-05 by repetitive element sequence-based PCR analysis in a pilot study of vaginal colonization. J Clin Microbiol. 2003 May;41(5):1881-7. doi: 10.1128/JCM.41.5.1881-1887.2003. PMID 12734221
- [Background] Sobel JD. Vaginitis in adult women. Obstet Gynecol Clin North Am. 1990 Dec;17(4):851-79. PMID 2092246
- [Background] Thomason JL, Gelbart SM, Scaglione NJ. Bacterial vaginosis: current review with indications for asymptomatic therapy. Am J Obstet Gynecol. 1991 Oct;165(4 Pt 2):1210-7. doi: 10.1016/s0002-9378(12)90729-2. PMID 1951577
- [Background] Pastore LM, Thorp JM Jr, Royce RA, Savitz DA, Jackson TP. Risk score for antenatal bacterial vaginosis: BV PIN points. J Perinatol. 2002 Mar;22(2):125-32. doi: 10.1038/sj.jp.7210654. PMID 11896517
- [Background] Kamara P, Hylton-Kong T, Brathwaite A, Del Rosario GR, Kristensen S, Patrick N, Weiss H, Figueroa PJ, Vermund SH, Jolly PE. Vaginal infections in pregnant women in Jamaica: prevalence and risk factors. Int J STD AIDS. 2000 Aug;11(8):516-20. doi: 10.1258/0956462001916425. PMID 10990336
- [Background] Gibney L, Macaluso M, Kirk K, Hassan MS, Schwebke J, Vermund SH, Choudhury P. Prevalence of infectious diseases in Bangladeshi women living adjacent to a truck stand: HIV/STD/hepatitis/genital tract infections. Sex Transm Infect. 2001 Oct;77(5):344-50. doi: 10.1136/sti.77.5.344. PMID 11588280
- [Background] Goldenberg RL, Klebanoff MA, Nugent R, Krohn MA, Hillier S, Andrews WW. Bacterial colonization of the vagina during pregnancy in four ethnic groups. Vaginal Infections and Prematurity Study Group. Am J Obstet Gynecol. 1996 May;174(5):1618-21. doi: 10.1016/s0002-9378(96)70617-8. PMID 9065140
- [Background] Sewankambo N, Gray RH, Wawer MJ, Paxton L, McNaim D, Wabwire-Mangen F, Serwadda D, Li C, Kiwanuka N, Hillier SL, Rabe L, Gaydos CA, Quinn TC, Konde-Lule J. HIV-1 infection associated with abnormal vaginal flora morphology and bacterial vaginosis. Lancet. 1997 Aug 23;350(9077):546-50. doi: 10.1016/s0140-6736(97)01063-5. PMID 9284776
- [Background] Allsworth JE, Peipert JF. Prevalence of bacterial vaginosis: 2001-2004 National Health and Nutrition Examination Survey data. Obstet Gynecol. 2007 Jan;109(1):114-20. doi: 10.1097/01.AOG.0000247627.84791.91. PMID 17197596
- [Background] Hay PE, Lamont RF, Taylor-Robinson D, Morgan DJ, Ison C, Pearson J. Abnormal bacterial colonisation of the genital tract and subsequent preterm delivery and late miscarriage. BMJ. 1994 Jan 29;308(6924):295-8. doi: 10.1136/bmj.308.6924.295. PMID 8124116
- [Background] Eschenbach DA. Bacterial vaginosis and anaerobes in obstetric-gynecologic infection. Clin Infect Dis. 1993 Jun;16 Suppl 4:S282-7. doi: 10.1093/clinids/16.supplement_4.s282. PMID 8324132
- [Background] Hawes SE, Hillier SL, Benedetti J, Stevens CE, Koutsky LA, Wolner-Hanssen P, Holmes KK. Hydrogen peroxide-producing lactobacilli and acquisition of vaginal infections. J Infect Dis. 1996 Nov;174(5):1058-63. doi: 10.1093/infdis/174.5.1058. PMID 8896509
- [Background] Puapermpoonsiri S, Kato N, Watanabe K, Ueno K, Chongsomchai C, Lumbiganon P. Vaginal microflora associated with bacterial vaginosis in Japanese and Thai pregnant women. Clin Infect Dis. 1996 Oct;23(4):748-52. doi: 10.1093/clinids/23.4.748. PMID 8909838
- [Background] Reid G, Burton J. Use of Lactobacillus to prevent infection by pathogenic bacteria. Microbes Infect. 2002 Mar;4(3):319-24. doi: 10.1016/s1286-4579(02)01544-7. PMID 11909742
- [Background] Hillier SL, Krohn MA, Klebanoff SJ, Eschenbach DA. The relationship of hydrogen peroxide-producing lactobacilli to bacterial vaginosis and genital microflora in pregnant women. Obstet Gynecol. 1992 Mar;79(3):369-73. doi: 10.1097/00006250-199203000-00008. PMID 1738516
- [Background] Avonts D, Sercu M, Heyerick P, Vandermeeren I, Meheus A, Piot P. Incidence of uncomplicated genital infections in women using oral contraception or an intrauterine device: a prospective study. Sex Transm Dis. 1990 Jan-Mar;17(1):23-9. PMID 2305333
- [Background] Soper DE, Bump RC, Hurt WG. Bacterial vaginosis and trichomoniasis vaginitis are risk factors for cuff cellulitis after abdominal hysterectomy. Am J Obstet Gynecol. 1990 Sep;163(3):1016-21; discussion 1021-3. doi: 10.1016/0002-9378(90)91115-s. PMID 2403128
- [Background] Bukusi EA, Cohen CR, Meier AS, Waiyaki PG, Nguti R, Njeri JN, Holmes KK. Bacterial vaginosis: risk factors among Kenyan women and their male partners. Sex Transm Dis. 2006 Jun;33(6):361-7. doi: 10.1097/01.olq.0000200551.07573.df. PMID 16547451
- [Background] Sexually transmitted diseases treatment guidelines 2002. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 May 10;51(RR-6):1-78. PMID 12184549
- [Background] Eschenbach DA, Hillier S, Critchlow C, Stevens C, DeRouen T, Holmes KK. Diagnosis and clinical manifestations of bacterial vaginosis. Am J Obstet Gynecol. 1988 Apr;158(4):819-28. doi: 10.1016/0002-9378(88)90078-6. PMID 3259075
- [Background] Hillier SL, Kiviat NB, Hawes SE, Hasselquist MB, Hanssen PW, Eschenbach DA, Holmes KK. Role of bacterial vaginosis-associated microorganisms in endometritis. Am J Obstet Gynecol. 1996 Aug;175(2):435-41. doi: 10.1016/s0002-9378(96)70158-8. PMID 8765265
- [Background] Larsson PG, Platz-Christensen JJ, Thejls H, Forsum U, Pahlson C. Incidence of pelvic inflammatory disease after first-trimester legal abortion in women with bacterial vaginosis after treatment with metronidazole: a double-blind, randomized study. Am J Obstet Gynecol. 1992 Jan;166(1 Pt 1):100-3. doi: 10.1016/0002-9378(92)91838-2. PMID 1733176
- [Background] Eschenbach DA. Bacterial vaginosis: emphasis on upper genital tract complications. Obstet Gynecol Clin North Am. 1989 Sep;16(3):593-610. PMID 2687747
- [Background] Watts DH, Krohn MA, Hillier SL, Eschenbach DA. Bacterial vaginosis as a risk factor for post-cesarean endometritis. Obstet Gynecol. 1990 Jan;75(1):52-8. PMID 2296423
- [Background] Newton ER, Prihoda TJ, Gibbs RS. A clinical and microbiologic analysis of risk factors for puerperal endometritis. Obstet Gynecol. 1990 Mar;75(3 Pt 1):402-6. PMID 2406660
- [Background] Paavonen J, Teisala K, Heinonen PK, Aine R, Laine S, Lehtinen M, Miettinen A, Punnonen R, Gronroos P. Microbiological and histopathological findings in acute pelvic inflammatory disease. Br J Obstet Gynaecol. 1987 May;94(5):454-60. doi: 10.1111/j.1471-0528.1987.tb03125.x. PMID 3580330
- [Background] Larsson PG, Platz-Christensen JJ, Forsum U, Pahlson C. Clue cells in predicting infections after abdominal hysterectomy. Obstet Gynecol. 1991 Mar;77(3):450-2. PMID 1992415
- [Background] Kurki T, Sivonen A, Renkonen OV, Savia E, Ylikorkala O. Bacterial vaginosis in early pregnancy and pregnancy outcome. Obstet Gynecol. 1992 Aug;80(2):173-7. PMID 1635726
- [Background] Riduan JM, Hillier SL, Utomo B, Wiknjosastro G, Linnan M, Kandun N. Bacterial vaginosis and prematurity in Indonesia: association in early and late pregnancy. Am J Obstet Gynecol. 1993 Jul;169(1):175-8. doi: 10.1016/0002-9378(93)90157-e. PMID 8333449
- [Background] Hillier SL, Nugent RP, Eschenbach DA, Krohn MA, Gibbs RS, Martin DH, Cotch MF, Edelman R, Pastorek JG 2nd, Rao AV, et al. Association between bacterial vaginosis and preterm delivery of a low-birth-weight infant. The Vaginal Infections and Prematurity Study Group. N Engl J Med. 1995 Dec 28;333(26):1737-42. doi: 10.1056/NEJM199512283332604. PMID 7491137
- [Background] Silver HM, Sperling RS, St Clair PJ, Gibbs RS. Evidence relating bacterial vaginosis to intraamniotic infection. Am J Obstet Gynecol. 1989 Sep;161(3):808-12. doi: 10.1016/0002-9378(89)90406-7. PMID 2782365
- [Background] Hillier SL, Martius J, Krohn M, Kiviat N, Holmes KK, Eschenbach DA. A case-control study of chorioamnionic infection and histologic chorioamnionitis in prematurity. N Engl J Med. 1988 Oct 13;319(15):972-8. doi: 10.1056/NEJM198810133191503. PMID 3262199
- [Background] Taha TE, Hoover DR, Dallabetta GA, Kumwenda NI, Mtimavalye LA, Yang LP, Liomba GN, Broadhead RL, Chiphangwi JD, Miotti PG. Bacterial vaginosis and disturbances of vaginal flora: association with increased acquisition of HIV. AIDS. 1998 Sep 10;12(13):1699-706. doi: 10.1097/00002030-199813000-00019. PMID 9764791
- [Background] Martin HL, Richardson BA, Nyange PM, Lavreys L, Hillier SL, Chohan B, Mandaliya K, Ndinya-Achola JO, Bwayo J, Kreiss J. Vaginal lactobacilli, microbial flora, and risk of human immunodeficiency virus type 1 and sexually transmitted disease acquisition. J Infect Dis. 1999 Dec;180(6):1863-8. doi: 10.1086/315127. PMID 10558942
- [Background] Myer L, Denny L, Telerant R, Souza Md, Wright TC Jr, Kuhn L. Bacterial vaginosis and susceptibility to HIV infection in South African women: a nested case-control study. J Infect Dis. 2005 Oct 15;192(8):1372-80. doi: 10.1086/462427. Epub 2005 Sep 9. PMID 16170754
- [Background] Hay P. Recurrent Bacterial Vaginosis. Curr Infect Dis Rep. 2000 Dec;2(6):506-512. doi: 10.1007/s11908-000-0053-5. PMID 11095900
- [Background] Bradshaw CS, Morton AN, Hocking J, Garland SM, Morris MB, Moss LM, Horvath LB, Kuzevska I, Fairley CK. High recurrence rates of bacterial vaginosis over the course of 12 months after oral metronidazole therapy and factors associated with recurrence. J Infect Dis. 2006 Jun 1;193(11):1478-86. doi: 10.1086/503780. Epub 2006 Apr 26. PMID 16652274
- [Background] Myer L, Kuhn L, Denny L, Wright TC Jr. Recurrence of symptomatic bacterial vaginosis 12 months after oral metronidazole therapy in HIV-positive and -negative women. J Infect Dis. 2006 Dec 15;194(12):1797-9. doi: 10.1086/509625. No abstract available. PMID 17109360
- [Background] Hughes VL, Hillier SL. Microbiologic characteristics of Lactobacillus products used for colonization of the vagina. Obstet Gynecol. 1990 Feb;75(2):244-8. PMID 2300352
- [Background] Chimura T, Funayama T, Murayama K, Numazaki M. [Ecological treatment of bacterial vaginosis]. Jpn J Antibiot. 1995 Mar;48(3):432-6. Japanese. PMID 7752457
- [Background] Fredricks DN, Fiedler TL, Thomas KK, Oakley BB, Marrazzo JM. Targeted PCR for detection of vaginal bacteria associated with bacterial vaginosis. J Clin Microbiol. 2007 Oct;45(10):3270-6. doi: 10.1128/JCM.01272-07. Epub 2007 Aug 8. PMID 17687006
- [Derived] Ngugi BM, Hemmerling A, Bukusi EA, Kikuvi G, Gikunju J, Shiboski S, Fredricks DN, Cohen CR. Effects of bacterial vaginosis-associated bacteria and sexual intercourse on vaginal colonization with the probiotic Lactobacillus crispatus CTV-05. Sex Transm Dis. 2011 Nov;38(11):1020-7. doi: 10.1097/OLQ.0b013e3182267ac4. PMID 21992977
- [Derived] Hemmerling A, Harrison W, Schroeder A, Park J, Korn A, Shiboski S, Foster-Rosales A, Cohen CR. Phase 2a study assessing colonization efficiency, safety, and acceptability of Lactobacillus crispatus CTV-05 in women with bacterial vaginosis. Sex Transm Dis. 2010 Dec;37(12):745-50. doi: 10.1097/OLQ.0b013e3181e50026. PMID 20644497